CLINICAL TRIAL: NCT03223688
Title: Effectiveness of Adjunctive Sensory Integration Therapy for Children With Developmental Delay in an Early Intervention Program
Brief Title: Early Intervention for Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Liang-Jen, Associate Professor and Visiting Staff, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105-1742C1
Record Dates: First submitted 2017-07-06; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Child Development; Developmental Delay; Early Intervention
MeSH Terms: conditions — Learning Disabilities | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Day-Care early intervention program (Experimental): The daily treatment session had eight children along with their major caregivers. The treatment was conducted by two experienced occupational therapists (OT), and each session lasted for four hours in the week-day morning with a 10-minute break. The goal of the sessions was to enhance children's development through cognitive training, behavioral modification plan and parenting skill training. Said therapists assisted the caregivers in improving their nurturing and parenting skills with their children, as well as their techniques with regards to influencing them.
  Interventions: Behavioral: Day-Care early intervention program
- OPD+SI intervention program (Experimental): The treatment program had eight children along with their major caregivers. The treatment was also performed by two experienced OT, and each session lasted for one hours, once a week. The sessions consisted of cognitive training, behavioral modification plan and parenting skill training. Adjunctive SI therapy was also performed by said OT for improving children's sensory motor development in an additional hour.
  Interventions: Behavioral: OPD+SI intervention program
- OPD intervention program (Active Comparator): The treatment program had eight children along with their major caregivers. The treatment was also performed by two experienced OT, and each session lasted for one hours, once a week. The sessions consisted of cognitive training, behavioral modification plan and parenting skill training.
  Interventions: Behavioral: OPD intervention program

INTERVENTIONS:
Behavioral: Day-Care early intervention program — The daily treatment session had eight children along with their major caregivers. The treatment was conducted by two experienced occupational therapists (OT), and each session lasted for four hours in the week-day morning with a 10-minute break. The goal of the sessions was to enhance children's development through cognitive training, behavioral modification plan and parenting skill training.
  Arms: Day-Care early intervention program
Behavioral: OPD+SI intervention program — The treatment program had eight children along with their major caregivers. The treatment was also performed by two experienced OT, and each session lasted for one hours, once a week. The sessions consisted of cognitive training, behavioral modification plan and parenting skill training. Adjunctive SI therapy was also performed by said OT for improving children's sensory motor development in an additional hour.
  Other Names: Adjunctive Sensory Integration (SI) Therapy
  Arms: OPD+SI intervention program
Behavioral: OPD intervention program — The treatment program had eight children along with their major caregivers. The treatment was also performed by two experienced OT, and each session lasted for one hours, once a week. The sessions consisted of cognitive training, behavioral modification plan and parenting skill training.
  Arms: OPD intervention program

SUMMARY:
This study aims to investigate the effectiveness of early intervention program in Department of Children and Adolescent Psychiatry, Kaohsiung Chang Gung Memorial Hospital. The investigators assume that the frequency of early-intervention and degree of family involvement will be associate with the treatment outcome.

DETAILED DESCRIPTION:
This prospective, non-randomized, open-label study is performed to assess the effects of adjunctive SI in the family-based treatment program of children with developmental delay (DD). The study subjects are children with DD who attended an early intervention (EI) program at Kaohsiung Chang Gung Memorial Hospital, which is the largest general hospital in the Southern Taiwan. Each participating child undergo a joint assessment by a pediatrician, a rehabilitation doctor, a child psychiatrist, a speech therapist, a physical therapist, an occupational therapist, and a social worker. Once the diagnosis of developmental delay is confirmed, the child will be scheduled for prescribed family-based early intervention in the same hospital. Children (between 2 to 4 years old) who attend the program will be enrolled in this study. Informed consent will be obtained from the children and their primary caregivers after they received a complete description of the study. The participants are categorized into three different groups based on their intervention method. The choice of intervention method will be according to the willingness and expedience of the children's caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children with Developmental Delay
* The caregivers are able to participate in the treatment program

Exclusion Criteria:

* Autism
* Cerebral palsy

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Changes of children's development | Assessment will be performed at baseline and 6-month after the baseline
  Mullen Scales of Early Learning

SECONDARY OUTCOMES:
Changes of caregivers' life quality | Assessment will be performed at baseline and 6-month after the baseline
  The World Health Organization Quality of Life- BREF (WHOQOL-BREF)
Changes of caregivers' parenting stress | Assessment will be performed at baseline and 6-month after the baseline
  The Parenting Stress Index-Short Form (PSI-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Jen Wang, Principal Investigator — Chang Gung Memorial Hospital, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No